CLINICAL TRIAL: NCT05336708
Title: The Effect of Acupressure on Fatigue in Nursing Students: A Randomized Controlled Study
Brief Title: The Effect of Acupressure on Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Esra Cavusoglu, Research assistant, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MersinUu
Record Dates: First submitted 2022-04-05; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Interventional
Keywords: Fatigue; Nursing students; Acupressure
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, two-arm, randomized controlled clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupressure group (Experimental): The acupressure (experimental) group will apply acupressure to themselves three times a week for a total of 12 sessions for four weeks.
  Interventions: Other: Acupressure Group
- Sham Acupressure Group (Sham Comparator): The sham acupressure group will apply acupressure to themselves three times a week for a total of 12 sessions for four weeks.
  Interventions: Other: Sham Acupressure Group

INTERVENTIONS:
Other: Acupressure Group — In the acupressure group, acupressure will be applied to the heart meridian 7th point (HT7), large intestine meridian 4th point (LI4), stomach meridian 36th point (ST36) and spleen meridian 6th point (SP6). After pressing each point for a certain period of time, a total of two minutes of rest periods will be applied by the researcher.
  Other Names: Experimental Group
  Arms: Acupressure group
Other: Sham Acupressure Group — In the sham acupressure group, acupressure will be applied on the bone region where the meridians do not pass, approximately 1-1.5 cm away from the HT7, LI4, ST36, SP6 points. The application process will continue in the same way with acupressure group and the pressure intensity will be less.
  Other Names: Sham Group
  Arms: Sham Acupressure Group

SUMMARY:
In this study, it is aimed to determine the effect of acupressure on fatigue in nursing students.

DETAILED DESCRIPTION:
In this study, 68 nursing students were randomly assigned to the acupressure and placebo (sham) acupressure groups. In the acupressure group (n=34), compression was applied to the 7th point of the heart meridian (HT7), the 4th point of the large intestine meridian (LI4), the 36th point of the stomach meridian (ST36), and the 6th point of the spleen meridian (SP6). Depending on the preparation and compression time at each point, the session duration of each student lasted an average of 20 minutes. In the sham group (n=34), pressure was applied approximately 1-1.5 cm away from the HT7, LI4, ST36, SP6 points. In the sham group, the acupressure application time lasted for an average of 20 minutes. At the end of the application, after the data collection process was completed, the sham group was taught the correct acupuncture points. Students applied acupressure three times a week for a total of 12 sessions for four weeks. Data were collected before and four weeks after the application in the acupressure and sham acupressure groups.

ELIGIBILITY:
Inclusion Criteria:

* Students studying at Mersin University Faculty of Nursing as 4th grade during the data collection date,
* Those who agree to participate in the study,
* No deformity or lesions in the areas where acupressure will be applied
* No acupressure experience
* No sleep disorder diagnosis and no medical treatment
* No diagnosis of anxiety disorder and no medical treatment No diagnosis of depression and no medical treatment
* Coffee, cigarette and alcohol-free,
* No mental illness,
* Able to understand and speak Turkish and
* Those who signed the Informed Consent Form will be included in the study.

Exclusion Criteria:

* Students studying at Mersin University Faculty of Nursing outside the 4th grade during the data collection date,
* Those who do not agree to participate in the study,
* Those who have any deformity or lesion in the areas where acupressure will be applied
* Experienced with acupressure
* Diagnosed with sleep disorder and receiving medical treatment
* Diagnosed with anxiety disorder and receiving medical treatment
* Diagnosed with depression and receiving medical treatment
* Coffee, cigarette and alcohol addiction,
* Having mental illness,
* who cannot understand or speak Turkish
* Those who do not sign the Informed Consent Form will not be included in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Fatigue evaluated using the Fatigue Severity Scale | Change from before implementation and 4th week of practice
  It is a Likert-type scale consisting of a total of nine items, each item being evaluated between 1 and 7 (1=I totally disagree, 7=I totally agree). The fatigue score is obtained by dividing the total score obtained from the scale by the number of scale items. The score that can be obtained from the scale varies between 9 and 63. A high score indicates an increased level of fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Meral Gün, Doctorate, Study Director — Mersin University
Locations (1):
- Mersin Üniversitesi, Mersin, Yenişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No